CLINICAL TRIAL: NCT00179218
Title: The Effects of Resistance Exercise and Protein Supplementation in Hemodialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Alp Ikizler, MD, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 50149; R01DK045604 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Dietary Supplements; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): only protein supplementation
  Interventions: Drug: nutritional supplementation
- 2 (Active Comparator): protein supplementation plus exercise
  Interventions: Drug: nutritional supplementation; Behavioral: exercise

INTERVENTIONS:
Drug: nutritional supplementation — oral administration of 2 cans of protein supplement (lactose-free formula that contains a total of 960 kilocalories: 132.8 kilocalories from protein, 412.8 kilocalories from carbohydrates, and 412.8 kilocalories from fat); every other day, 3 days per week, for 6 months
Behavioral: exercise — leg press exercise; every other day, 3 days per week, for 6 months
  Arms: 2

SUMMARY:
The objective of this study is to determine how protein supplementation, with or without exercise, affects functional capacity, strength, body composition, and physical activity in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* On hemodialysis for more than 3 months, on a thrice weekly hemodialysis program;
* Adequately dialyzed (Kt/V ≥ 1.2).
* Age ≥ 18 years old.

Exclusion Criteria:

* Patients unable to perform exercise due to cardiovascular disease, osteoarthritis, etc., as determined by the PI and the primary physician of the subject.
* Pregnant women.
* Patients hospitalized within the last month prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-04; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
increase in lean body mass | 12 months

SECONDARY OUTCOMES:
increase in physical functioning | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States